CLINICAL TRIAL: NCT03242265
Title: Open Label, Prospective, Cross-Sectional Clinical Performance Study of the in Vitro Diagnostic Device NK VueTM: Measurement of Natural Killer Cell Activity in Whole Blood in Men Being Screened for Prostate Cancer With Biopsy
Brief Title: Measurement of Natural Killer Cell Activity in Whole Blood in Men Being Screened for Prostate Cancer With Biopsy
Acronym: ANKA-PCA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: ATGen Canada Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: ANKA-PCA
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Immunity, Innate; Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: NK cell activity not provided to investigator prior to biopsy; results of biopsy not provided to biochemistry lab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: IVDD for NK cell activity in whole blood — Two samples of one mL of blood (for baseline IFN-gamma activity and for NK cell activity) and blood samples collected for C-Reactive Protein and White Blood Cell Count, taken up to 8 weeks prior to biopsy and before treatment with antibiotics.
  Other Names: NK Vue

SUMMARY:
This study will look at measuring the activity of natural killer (NK) cells using the in vitro diagnostic device NK Vue in subjects being screened for prostate cancer using prostate biopsy.

DETAILED DESCRIPTION:
The NK Vue diagnostic test for natural killer cell activity uses the principle of stimulation of whole blood with a proprietary cytokine followed by the quantitative detection of interferon-gamma using an immunoassay. NK Vue is intended to be used for the monitoring of the immune status of individuals. Measurement of NK cell activity could be a useful tool for assessing changes in immunosurveillance in patients with conditions or diseases where NK cell activity has been shown to be affected.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged ≥ 18 years old
2. Able to read and sign an approved informed consent form
3. Soon to be undergoing a needle prostate biopsy for suspected prostate cancer; patients with a history of prior biopsy are not excluded provided the biopsy was negative
4. All prior and current recorded PSA levels are < 11 ng/mL (minimum of 2 values must be available)
5. Digital Rectal Exam performed or scheduled to be performed prior to biopsy

Exclusion Criteria:

1. Any other established malignancy with the exception of basal cell carcinoma
2. At time of blood collection, an active infection (eg bacterial, viral etc.) as declared by the patient
3. Chronic inflammatory condition requiring anti-inflammatory treatment such as rheumatoid arthritis, Crohn's or ulcerative colitis, Lupus or any connective tissue condition which, in the opinion of the investigator, might affect the immune response
4. Presently taking any of the following classes of medications on a regular basis:

   * 5-alpha reductase inhibitors
   * Anti-inflammatories, with the exception of low dose (81 mg) acetylsalicylic acid
   * Anti-androgens
   * Testosterone replacement therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-representation (must have a prostate gland)
Enrollment: 84 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
The ability of NK cell activity to predict prostate cancer (yes/no) on biopsy | NK cell activity is measured up to 8 weeks prior to biopsy and prior to starting any antibiotic treatment
  Test performance of NK Vue will be assessed by logistic regression, both unadjusted and adjusted for the effects of at least PSA, age, digital rectal examination, and family history

SECONDARY OUTCOMES:
The ability of NK cell activity to predict tumor grade (Gleason 2-6 vs. no cancer; Gleason 7-10 vs. no cancer) | NK cell activity is measured up to 8 weeks prior to biopsy and prior to starting any antibiotic treatment
  Test performance of NK Vue will be assessed by multinomial logistic regression, using the following known predictors of prostate cancer: age, ethnicity, PSA history, family history of prostate cancer, prostate volume, digital rectal examination findings, and number of prior biopsies.
Test performance metrics of NK Vue and PSA (each alone) | NK cell activity is measured up to 8 weeks prior to biopsy and prior to starting any antibiotic treatment
  The sensitivity, specificity, positive and negative predictive values for the detection of prostate cancer, will be calculated using Receiver Operating Characteristics analysis (at a cut-off of 4 ng/mL for PSA and at a cut-off of 200 pg/mL for NK Vue). Other cut-offs may be used to perform additional statistical analyses for test performance.
Impact of combination of NK Vue and PSA on the test performance of PSA | NK cell activity is measured up to 8 weeks prior to biopsy and prior to starting any antibiotic treatment
  The sensitivity, specificity, positive and negative predictive values for the detection of prostate cancer, will be calculated using Receiver Operating Characteristics analysis under combined conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Neil E Fleshner, MPH,MD,FRCSC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Center, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barkin J, Rodriguez-Suarez R, Betito K. Association between natural killer cell activity and prostate cancer: a pilot study. Can J Urol. 2017 Apr;24(2):8708-8713. PMID 28436356
- [Background] Koo KC, Shim DH, Yang CM, Lee SB, Kim SM, Shin TY, Kim KH, Yoon HG, Rha KH, Lee JM, Hong SJ. Reduction of the CD16(-)CD56bright NK cell subset precedes NK cell dysfunction in prostate cancer. PLoS One. 2013 Nov 4;8(11):e78049. doi: 10.1371/journal.pone.0078049. eCollection 2013. PMID 24223759